CLINICAL TRIAL: NCT05347979
Title: An Open-Label, Drug-Drug Interaction Study Designed to Evaluate the Effect of Relacorilant on the Pharmacokinetics of the Sensitive P-glycoprotein Substrate Dabigatran Etexilate in Healthy Subjects
Brief Title: Effect of Relacorilant on the Pharmacokinetics of the Sensitive P-glycoprotein Substrate Dabigatran Etexilate in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CORT125134-132
Record Dates: First submitted 2022-04-18; First posted 2022-04-27 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Cushing Syndrome; Neoplasms
MeSH Terms: conditions — Cushing Syndrome; Neoplasms | interventions — Dabigatran; relacorilant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dabigatran Etexilate (NIMP) and Relacorilant (IMP) (Experimental): Following an overnight fast, participants will receive 75 mg dabigatran etexilate on Day 1, 400 mg dose of relacorilant QD on Days 3 to 13, and 75 mg dabigatran etexilate on Day 12. On Day 12, dabigatran etexilate will be dosed at approximately the same time as the relacorilant dose.
  Interventions: Drug: Dabigatran Etexilate; Drug: Relacorilant

INTERVENTIONS:
Drug: Dabigatran Etexilate — Dabigatran will be administered orally as a 75 mg capsule on Day 1 and Day 12.
  Other Names: Pradaxa®
Drug: Relacorilant — Relacorilant will be administered orally as 4 X 100 mg capsules (400 mg) on Days 3 through 13.

SUMMARY:
The primary objective is to determine the effect of relacorilant on the pharmacokinetics (PK) of the sensitive P-glycoprotein (P-gp) substrate dabigatran etexilate.

DETAILED DESCRIPTION:
The investigational medicinal product (IMP), relacorilant, and the non-investigational medicinal product (NIMP), dabigatran etexilate, will be used to evaluate the effect of relacorilant on the PK of the sensitive P-gp substrate, dabigatran etexilate in healthy participants. Participants will receive a single dose of dabigatran etexilate before and after administration of daily (QD) doses of relacorilant for 11 days. As all participants will receive the same treatments, the study will be open-label and no randomization is required.

ELIGIBILITY:
Inclusion Criteria:

* Must agree to use an adequate method of contraception
* Healthy men or non-pregnant, non-lactating healthy women of non-childbearing potential
* Body mass index (BMI) of 19.0 to 32.0 kg/m^2 as measured at screening
* Weight ≥50 kg at screening

Exclusion Criteria:

* Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
* Presence or history of clinically significant allergy requiring treatment, as judged by the Investigator.
* Significant serious skin disease, including rash, food allergy, eczema, psoriasis, or urticaria
* History of clinically significant cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal disease, bleeding disorder or abnormal bleeding, or clinically significant active bleeding, congenital or acquired clotting disorders, neurological or psychiatric disorder
* History of esophagitis, gastritis, gastroesophageal reflux surgery, or significant trauma or surgery within 1 month of IMP/NIMP administration
* Have poor venous access that limits phlebotomy
* Evidence of current severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection
* Clinically significant abnormal clinical chemistry, hematology or thrombocytopenia, coagulation or urinalysis
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) antibody results
* Evidence of renal impairment at screening
* Pregnant or lactating women
* Women of childbearing potential. A woman is considered of childbearing potential unless she is permanently sterile or is postmenopausal
* Participants who have received any IMP in a clinical research study within 5 half-lives or within 30 days prior to first dose.
* Participants who are taking, or have taken, any prescribed or over-the-counter drug or herbal remedies in the 14 days before IMP/NIMP administration.
* Participants who are currently using glucocorticoids or have a history of systemic glucocorticoid use at any dose within the last 12 months before IMP/NIMP administration, or 3 months for inhaled products
* Participants who are taking, or have taken, heparin, vitamin K antagonists or anti-platelet agents within 1 month before IMP/NIMP administration
* Participants who are taking, or have taken, selective serotonin re-uptake inhibitors, serotonin and norepinephrine re-uptake inhibitors within 3 months before IMP/NIMP administration
* History of any drug or alcohol abuse in the past 2 years
* A confirmed positive alcohol urine test at screening or admission
* Current smokers and those who have smoked within the last 12 months
* Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months
* Positive drugs of abuse test result
* Male participants with pregnant or lactating partners
* Donation of blood within 2 months or donation of plasma within 7 days prior to first dose of study medication

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2022-07-19 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Dabigatran When Administered With and Without Relacorilant | Up to Day 14
Area Under the Curve from Time 0 to the Time of Last Measurable Concentration (AUC0-last) of Dabigatran When Administered With and Without Relacorilant | Up to Day 14
Area Under the Curve from Time 0 Extrapolated to Infinity (AUC 0-inf) of Dabigatran When Administered With and Without Relacorilant | Up to Day 14

SECONDARY OUTCOMES:
Plasma Concentrations of Relacorilant | Up to Day 6
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 30 days post final dose
Number of Participants with Clinically Significant Abnormalities in Blood Pressure and Heart Rate | Up to Day 14
Number of Participants with Clinically Significant Abnormalities in Electrocardiogram (ECG) Measurements | Up to Day 14
Number of Participants with Clinically Significant Abnormalities in Laboratory Safety Tests (Clinical Chemistry, Hematology, Urinalysis) | Up to Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Custodio, PhD, Study Director — Corcept Therapeutics
Locations (1):
- Site 01, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No